CLINICAL TRIAL: NCT04545190
Title: RibOSE - Effects of Glucose Ingestion During Resistance Exercise Training on Ribosomal Biogenesis in Skeletal Muscle
Brief Title: RibOSE - Glucose and Resistance Exercise Training
Acronym: RibOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Anne Sofie Lofthus, Administrator, Inland Norway University of Applied Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Trainome#024_2020
Record Dates: First submitted 2020-08-24; First posted 2020-09-10 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Strength/resistance training; Glucose supplementation; Skeletal muscle
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a 12-day placebo-controlled randomized clinical trial. Each day will consist of concomitant dietary intervention and resistance training. The dietary intervention consists of alternating days of ingesting glucose (GLU, 90 g) or placebo (PLAC) in connection with training. Likewise, training consists of alternating days of resistance training of the two legs (using identical training protocols), with Day 1 involving training of the first leg, Day 2 involving training of the second leg, Day 3 involving training of the first leg, etc. In this way, each of the two dietary interventions will be associated with training of one particular leg, allowing within-subject comparisons of the effects of GLU vs PLAC on muscle biology and recovery.
Who Masked: Participant, Investigator
Masking Description: On each intervention day, participants will receive boluses of supplements in accordance with his or her study ID number. The list that links this ID number to the randomization code will be kept with the person who generated the randomization code (and stored on a safe server) until completion of data sampling and cleaning of data on main outcome measures. The person resonsible for generating the randomization code will not be involved in any aspects of data sampling or handling. None of the project collaborators/participants will have access to this list during the intervention or during data handling.
  Half the participants (n=10) will commence the intervention with GLU on Day 1, while the other half will commence with PLAC (randomized). For participants starting with GLU, half will perform training on their dominant leg, while the other half will perform training on their non-dominant leg. The same will be the case for participants starting with PLAC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose (Active Comparator): Glucose will be ingested at three time points during resistance training (RT): 30 min prior to RT (30 g glucose mixed with 300 ml sugar-free Fun light lemonade), immediately prior to RT (30 g, 300 ml), and immediately after completion of training (30 g, 300 ml).
  Protein supplement will be ingested at two time points: 2 hours prior to RT (e.g. at 0700 hrs, 25 g) and immediately after completion of training (25 g).
  Placebo will be ingested during the afternoon (i.e. not during training; between 1800 hrs and 1900 hrs): 3 x 100 mg Stevia powder mixed with 3 x 300 ml sugar-free Fun light lemonade.
  (The dietary intervention spans from 2200 hrs on the evening prior to RT sessions to ~2.5 hrs after completion of RT. During this time frame, participants will ingest glucose and protein supplements only)
  Interventions: Dietary Supplement: Glucose
- Placebo (Placebo Comparator): Placebo will be ingested at three time points during resistance training (RT): 30 min prior to RT (100 mg Stevia powder mixed with 300 ml sugar-free Fun light lemonade), immediately prior to RT (100 mg, 300 ml), and immediately after completion of training (100 mg, 300 ml).
  Protein supplement will be ingested at two time points: 2 hours prior to RT (e.g. at 0700 hrs, 25 g) and immediately after completion of training (25 g).
  Glucose will be ingested during the afternoon (i.e. not during training; between 1800 hrs and 1900 hrs): 3 x 30 g glucose mixed with 3 x 300 ml sugar-free Fun light lemonade.
  (The dietary intervention spans from 2200 hrs on the evening prior to RT sessions to ~2.5 hrs after completion of RT. I.e.: during this period, participants will ingest placebo and protein supplements only)
  Interventions: Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Glucose — To investigate the effects of glucose intake during resistance training on muscle biological adaptations

SUMMARY:
The aim of the study is to investigate the effects of ingesting glucose during five bouts of resistance exercise on muscle biological charateristics in m. vastus lateralis of moderately trained healthy individuals (20-45 years of age, n=20)

DETAILED DESCRIPTION:
Muscular responses to resistance training vary extensively between humans, with many showing impaired growth. In such individuals, cellular plasticity is compromised, leading to reduced functional and health-beneficial outcomes of training. While this is likely due to a range of determinants, including epigenetic, genetic and physiological variables, recent studies suggest that it involves reduced ability to produce novel ribosomes in response to training. This eventually leads to less pronounced increases in protein synthesis, and thus decreased growth rates, and makes ribosomal content in muscle a potential proxy marker for training-associated muscle hypertrophy.

In a recent study, the investigators showed that increased resistance training volume was associated with more pronounced muscle growth, a trait that was associated with increased ribosomal biogenesis. Despite this, ~50 % of the participants did not exhibit true beneficial effects of increased training volume, which in turn coincided with reduced abilities to accumulate ribosomes. In such individuals, other means are likely necessary to circumvent the negative influence of genetic and epigenetic predispositions on muscle plasticity. Nutrient supplementation stand out as a potential therapy. However, at present, knowledge with regard to this perspective is limited to a selected few nutrients, with protein ingestion being the best studied potential adjuvant, for which adequate intake seems to be essential for achieving optimal muscle growth, potentially being interconnected with ribosomal synthesis. For other nutrients, such as glucose, little is know about their importance for muscle plasticity and ribosomal biogenesis.

In cell types such as cultivated kidney cells, exposure to high levels of glucose is an efficient mean to increase ribosomal biogenesis (and growth rates). This suggests that glucose is an important signaling molecule for increasing ribosomal production per se, perhaps acting as a ligand for signaling proteins or by acting to increase energy availability. In the human body (as opposed to cultured cells), glucose may also exert growth-stimulating effects by increasing insulin levels in blood. Overall, it thus seems plausible that glucose intake during resistance training may stimulate ribosomal biogenesis, in turn having beneficial effects for protein synthesis and muscle plasticity, perhaps acting in an additive manner to protein supplementation. At present, we do not know if this is the case, though studies have suggested that glucose ingestion during acute resistance training sessions may reduce training-induced muscle damage without affecting within-session work output (i.e. volume). This lack of knowledge is surprising given the long-standing appreciation of the beneficial effects of glucose intake for endurance performance, acting to delay muscular fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Moderately trained (i.e. having performed 2-8 resistance training sessions per 14 days for the last six months)

Exclusion Criteria:

* Not able to understand Norwegian
* Unstable cardiovascular disease
* Illness or injury contradicting heavy strength training
* Disabling musculoskeletal disease
* Serious mental illness
* Allergy to local anaesthesia
* Impaired glucose tolerance

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Total RNA in muscle tissue | Before the intervention and immediately after the intervention (i.e. after 5 training sessions of each leg)
  Total RNA content in m. vastus lateralis (ug per mg tissue)

SECONDARY OUTCOMES:
Ribosomal RNA in skeletal muscle | Before the intervention and immediately after the intervention (i.e. after 5 training sessions of each leg)
  Abundances of ribosomal RNA species in m. vastus lateralis measured using qPCR
Protein in skeletal muscle | Before the intervention and immediately after the intervention (i.e. after 5 training sessions of each leg)
  Abundances of protein species in m. vastus lateralis measured using Western blotting (e.g. ECM proteins)
Gene expression in skeletal muscle | Before the intervention and immediately after the intervention (i.e. after 5 training sessions of each leg)
  Abundances of mRNA species in m. vastus lateralis measured using qPCR
Muscle fractional synthesis rate | Immediately after the intervention
  Protein synthesis rate measured using heavy water (deuterium) and chromatography/spectrometry
Glucose in blood, after glucose/placebo intake | Immediately before glucose/placebo intake and 30 min, 45 min, 60 min and 195 min after initial glucose/placebo intake
  Glucose concentrations in blood (area under the curve), measured before and after intake of glucose/placebo on the two final days of the intervention (one day = glucose; one day = placebo)
Glucose in blood (after protein intake) | Immediately before protein intake and 45 min and 90 min after protein intake
  Glucose concentrations in blood (area under the curve), measured before and after intake of protein on the two final days of the intervention
Hormone concentrations in blood (after glucose/placebo intake) | Immediately before glucose/placebo intake and 30 min and 60 min after the initial glucose/placebo intake
  Abundances of insulin, c-peptide, testosterone, growth hormone, cortisol and inflammatory markers in blood (area under the curve), measured before and after intake of glucose/placebo on the two final days of the intervention (one day = glucose; one day = placebo)
Hormone concentrations in blood (after protein intake) | Immediately before protein intake and 90 min after protein intake
  Abundances of insulin, c-peptide, testosterone, growth hormone, cortisol and inflammatory markers in blood, measured after intake of protein on the two final days of the intervention
Unilateral lower body isokinetic muscle strength (during the intervention) | Before the intervention and after the second, fourth and sixth training session
  The ability of the knee extensors to exert maximal force during isokinetic movements (recovery/strength), measured before the intervention and at three time points during the intervention (~24 hours after training sessions)
Unilateral lower body isokinetic muscle strength (last days of the intervention) | Before the last training session and 30 min, 120 min and 24 hours after the last training session
  The ability of the knee extensors to exert maximal force during isokinetic movements (recovery/strength), measured before and at three time points after the last two training sessions (one day = glucose; one day = placebo)
Unilateral lower body isometric muscle strength (during the intervention) | Before the intervention and after the second, fourth and sixth training session
  The ability of the knee extensors to exert maximal force during isometric actions (recovery/strength), measured before the intervention and at three time points during the intervention (~24 hours after training sessions)
Unilateral lower body isometric muscle strength (last days of the intervention) | Before the last training session and 30 min, 120 min and 24 hours after the last training session
  The ability of the knee extensors to exert maximal force during isometric actions (recovery/strength), measured before and at three time points after the last two training sessions (one day = glucose; one day = placebo)
Perceived muscle soreness (during the intervention) | Before the intervention and 24 hours after each training session
  Muscular soreness measured before the intervention and at three time points during the intervention (~24 hours after training sessions) using a VAS-scale from 0 to 10 (0 = no soreness; 10 = maximal soreness)
Perceived feeling of the legs (during the intervention) | 30 min after each training session
  Feeling of the legs measured immediately after each training session using a 9-point scale (1 = very very good, 9 = very very heavy)

OTHER OUTCOMES:
Training diary | During each training session of the intervention
  Training volume (total kg lifted) during each day of the intervention
Body mass composition | Prior to the intervention
  Body mass composition measured using DXA
Dietary registration | During each day of the intervention
  Nutritional intake during each day of the intervention, tracked using MyFitnessPal
Unilateral lower body maximal strength | Before the intervention
  The ability of muscles of the lower body to exert maximal force during dynamic movements
Blind test glucose vs placebo comparators | Immediately after the intervention
  The ability to discriminate between glucose and placebo beverages, tested after the training intervention using a blinded randomized design: each participant will ingest six beverages (3 x glucose and 3 x placebo) and will be asked to identify theam as either glucose or placebo. The "ability to discriminate" will be determined based on analyses of the full study population
Deuterium in spit | On each day of the intervention
  Deuterium levels in spit on each day during the intervention measured using chromatography/spectrometry (sampled prior to each training session)
Fasting blood glucose | Before the intervention and immediately after the intervention
  Fasting blood glucose measured in serum, measured before the intervention and prior to training on the last two days of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stian Ellefsen, PhD, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammarstrom D, Ofsteng S, Koll L, Hanestadhaugen M, Hollan I, Apro W, Whist JE, Blomstrand E, Ronnestad BR, Ellefsen S. Benefits of higher resistance-training volume are related to ribosome biogenesis. J Physiol. 2020 Feb;598(3):543-565. doi: 10.1113/JP278455. Epub 2020 Jan 15. PMID 31813190